CLINICAL TRIAL: NCT02963311
Title: An Open-Label, Single-Arm, Multicenter Pilot Study to Evaluate Safety, Tolerability, and Efficacy of ALN-PCSSC in Subjects With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: A Study of ALN-PCSSC in Participants With Homozygous Familial Hypercholesterolemia (HoFH)
Acronym: ORION-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-PCS-16-02
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — ALN-PCS; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALN-PCSSC (Experimental): 300 milligrams (mg) administered subcutaneous (SC) on Day 1. Participants with a mean serum proprotein convertase subtilisin/kexin type 9 (PCSK9) levels not suppressed by >70% at Day 60 or Day 90, as compared to baseline, will receive a second dose at Day 90 or Day 104, respectively, based on PCSK9 levels from the previous visit. Participants also received standard of care as background therapy.
  Interventions: Drug: ALN-PCSSC; Drug: Standard of Care

INTERVENTIONS:
Drug: ALN-PCSSC — ALN-PCSSC is a small interfering ribonucleic acid (siRNA) that inhibits PCSK9 synthesis and is given as SC injections.
  Other Names: PCSK9 synthesis inhibitor
Drug: Standard of Care — Included maximally-tolerated statin therapy and/or other low density lipoprotein-cholesterol (LDL-C)-lowering therapies.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of ALN-PCSSC in participants with homozygous familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥12 years of age with a diagnosis of homozygous familial hypercholesterolemia by genetic confirmation or a clinical diagnosis based on a history of an untreated low-density lipoprotein cholesterol (LDL-C) concentration >500 mg/deciliter (dL) [13 millimoles/liter (mmol/L)] together with either xanthoma before 10 years of age or evidence of heterozygous familial hypercholesterolemia in both parents.
* Stable on a low-fat diet.
* Stable on pre-existing, lipid-lowering therapies (such as statins, cholesterolabsorption inhibitors, bile-acid sequestrants, or combinations thereof) for at least 4 weeks with no planned medication or dose change for the duration of study participation.
* Fasting central lab LDL-C concentration >130 mg/dL (3.4 mmol/L) and triglyceride concentration <400 mg/dL (4.5 mmol/L).
* Body weight of 40 kilograms (kg) or greater at screening.

Exclusion Criteria:

* LDL or plasma apheresis within 8 weeks prior to the screening visit, and no plan to receive it during the study because of the attendant difficulty in maintaining stable concentrations of LDL-C while receiving apheresis.
* Use of mipomersen or lomitapide therapy within 5 months of screening.
* Previous treatment with monoclonal antibodies directed towards PCSK9 within 8 weeks of screening.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kees Hovingh, MD, PhD, Principal Investigator — Department of Vascular Medicine, Academic Medical Center
Locations (3):
- Research Site 201001, Los Angeles, California, United States
- Research Site 231001, Amsterdam, Netherlands
- Research Site 227001, Parktown, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Inclisiran: 300 milligrams (mg) administered subcutaneous (SC) on Day 1. Participants with a mean serum proprotein convertase subtilisin/kexin type 9 (PCSK9) levels not suppressed by >70% at Day 60 or Day 90, as compared to baseline, will receive a second dose at Day 90 or Day 104, respectively, based on PCSK9 levels from the previous visit. Participants also received standard of care as background therapy.
  Inclisiran: Inclisiran is a small interfering ribonucleic acid (siRNA) that inhibits PCSK9 synthesis and is given as SC injections.
  Standard of Care: Included maximally-tolerated statin therapy and/or other low density lipoprotein-cholesterol (LDL-C)-lowering therapies.
Period: Overall Study
Arm/Group | Inclisiran
Started | 9
Completed | 4
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 4

BASELINE CHARACTERISTICS:
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 1
  South Africa | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Day 1 to Day 90 in LDL-C
Description: Due to the small number of subjects, and the fact that the data are not normally distributed, the data are presented as descriptive statistics with no inferential and limited summary statistics presented.
Time Frame: Day 1, Day 90
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change | -12.26 [-43.75 to 19.24]

2. Primary Outcome: Percentage Change From Day 1 to Day 180 (or Final Visit) in LDL-C
Time Frame: Day 1, Day 180 (or Final Visit)
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change | -20.96 [-49.97 to 8.05]

3. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in LDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -56.3 (115.18)
  Day 180 | -105.3 (116.44)

4. Secondary Outcome: Percentage Change From Day 1 to Day 60 and to Day 90 in PCSK9
Time Frame: Day 1, Day 60, Day 90
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 60 | -64.9 (18.33)
  Day 90 | -59.0 (16.46)

5. Secondary Outcome: Absolute Change From Day 1 to Day 60 and to Day 90 in PCSK9
Time Frame: Day 1, Day 60, Day 90
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
ng/mL
  Day 60 | -654.1 (564.67)
  Day 90 | -602.3 (559.61)

6. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Total Cholesterol
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -13.9 (14.84)
  Day 180 | -19.8 (13.68)

7. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Total Cholesterol
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -77.8 (103.41)
  Day 180 | -118.0 (103.52)

8. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Triglycerides
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -21.0 (30.99)
  Day 180 | -20.13 (11.67)

9. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Triglycerides
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -35.5 (38.76)
  Day 180 | -26.3 (24.64)

10. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in HDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -12.1 (17.98)
  Day 180 | -19.8 (11.78)

11. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in HDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -6.0 (9.13)
  Day 180 | -9.5 (4.73)

12. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Non-HDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -13.9 (14.78)
  Day 180 | -19.7 (13.93)

13. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Non-HDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -71.8 (97.70)
  Day 180 | -108.5 (99.38)

14. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in VLDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | 8.5 (65.28)
  Day 180 | 55.5 (131.92)

15. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in VLDL-C
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -15.5 (28.41)
  Day 180 | -3.3 (37.32)

16. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Apolipoprotein A1
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -8.3 (12.95)
  Day 180 | -14.2 (14.44)

17. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Apolipoprotein A1
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -11.5 (17.52)
  Day 180 | -19.8 (19.00)

18. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Apolipoprotein B
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -26.6 (14.98)
  Day 180 | -25.0 (14.50)

19. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Apolipoprotein B
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
mg/dL
  Day 90 | -95.3 (78.16)
  Day 180 | -86.3 (72.02)

20. Secondary Outcome: Percentage Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Lipoprotein-a
Description: The reported percent change value is the per participant calculated Mean.
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
percent change
  Day 90 | -3.5 (15.70)
  Day 180 | -11.8 (15.15)

21. Secondary Outcome: Absolute Change From Day 1 to Day 90 and to Day 180 (or Final Visit) in Lipoprotein-a
Time Frame: Day 1, Day 90, Day 180 (or Final Visit)
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Inclisiran
Number analyzed (Participants) | 4
nmol/L
  Day 90 | 13.5 (21.92)
  Day 180 | -23.8 (52.73)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Inclisiran
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inclisiran (N=4)
Angina unstable (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=4)
Angina unstable (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cystitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT02963311/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02963311/SAP_001.pdf